CLINICAL TRIAL: NCT01501058
Title: Parent-Assisted Social Skill Training Program in the Adolescents With Autism Spectrum Disorder
Brief Title: Parent-supported Social Skills Training for Teens With Autism Spectrum Disorders (PEERS-K)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PEERSK2011
Record Dates: First submitted 2011-12-19; First posted 2011-12-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

ARMS (2):
- case group (Experimental)
  Interventions: Behavioral: parent-assisted social skills training program for adolescents with autism spectrum disorder
- waitlist control group (Other): For this group, same intervention with the Experimental group will be provided after waiting for 14 weeks.
  Interventions: Behavioral: Delayed intervention

INTERVENTIONS:
Behavioral: parent-assisted social skills training program for adolescents with autism spectrum disorder — The subjects will participate in the treatment program weekly for a total of 14 weeks. The final visit will be made at the point three months after the completion of treatment to see mid- and long-term effects.
  Arms: case group
Behavioral: Delayed intervention — Intervention is provided to Waitlist Control Group after waiting for 14 weeks
  Arms: waitlist control group

SUMMARY:
This study aims to develop a parent-assisted social skills training program for adolescents with autism spectrum disorder(ASD) and verify therapeutic effects of the program through case-control study.

1. Both the case and the control of this study shall be a high-functioning group consisting of adolescents aged 11 to 18 years with ASD and an IQ of 80 or over. A total of 40 adolescents will be recruited and divided into two groups of twenty. One will be the case group and the other will be the waitlist control group. Again, the case will be divided into two sub-groups of ten and carry out this new developed program for both parents and adolescents. That is, the program will be carried out two times in each of both groups. The waitlist control group will be allowed to receive personal outpatient treatment and general therapeutic intervention from community while waiting.
2. Effects of the program will be measured both at the case and the control by using a scale which measures social interaction, quality of peer relationship, disposition of autism and social anxiety. Equal assessments for both the case and the control will be conducted right before the beginning of the program and right after the completion of the program and some of the survey will be retried in order to see mid- and long-term effects three months after the completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* 11 to 18 years with ASD and an IQ of 65 or over

Exclusion Criteria:

* Adolescents who are hard to understand the content of treatment and carry out the task due to their IQs or limited linguistic abilities
* Adolescents who are uncooperative in the treatment, lack motives and are hard to participate voluntarily
* Adolescents who have behavior problems so clinically significant that they affects the therapeutic procedure or problems in controlling their emotion

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Test of Adolescent Social Skills Knowledge(TASSK) at 3month | baseline,3month
  The TASSK is a 22-item criterion-referenced test developed for this study to assess the teen's knowledge about the specific social skills taught during the intervention. Two items were derived from key elements of each of the 11 didactic lessons. Teens were presented with sentence stems and asked to choose the best option from two possible answers. Scores range from 0 to 22, with higher scores reflecting greater knowledge of teen social skills.

SECONDARY OUTCOMES:
Change from baseline in Social Skills Rating Scale (SSRS) at 3 month | baseline,3month
  The SSRS consists of 38-items and took approximately 10 min to complete. Questionnaires were completed independently by the teen's parent and teacher. For example, items included ''Starts conversations rather than waiting for someone to talk first.'' The items were rated as either ''Never,'' ''Sometimes,'' or ''Very Often.'' The Social Skills and Problem Behaviors scales were derived from factor analysis.
Change from baseline in Friendship Qualities Scale (FQS) at 3month | baseline,3month
  The FQS is a teen self-report measure that assesses the quality of best friendships. It consists of 23 yes/no questions from five different subscales (Companionship, Closeness, Help, Security, and Conflict) and took approximately 10 min to complete. Teens were instructed to identify their best friend and keep this friendship in mind while completing this measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea